CLINICAL TRIAL: NCT00156065
Title: A Multicenter, Randomized, Double-Blind, Flexible-Dose, Long-Term Extension Trial of the Safety and Maintenance of Effect of Asenapine Using Haloperidol Positive Control in Subjects Who Complete Protocol 041023 [NCT00156104]
Brief Title: Long-Term Efficacy and Safety of Asenapine Using Haloperidol as a Positive Control (41513)(COMPLETED)(P05785)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05785; Hera;; 41513
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2010-04-07 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Haloperidol; asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Haloperidol/Haloperidol (Active Comparator): Haloperidol in original study (NCT00156104) and in current long-term extension.
  Interventions: Drug: Haloperidol
- Asenapine/Asenapine (Experimental): Asenapine in original study and asenapine in current long-term extension.
  Interventions: Drug: Asenapine
- Placebo/Asenapine (Experimental): Double-Blind subjects randomized to only placebo medication for 6 weeks in the short-term 041023 asenapine trial, were randomized (double-blind) into the long-term 041513 asenapine extension trial and received asenapine 5 mg BID for Week 1. After Week 1, subjects received asenapine (either 5 mg BID or 10 mg BID) for the remainder of the 52-week trial.
  Interventions: Drug: Asenapine

INTERVENTIONS:
Drug: Haloperidol — 2-8 mg BID
  Arms: Haloperidol/Haloperidol
Drug: Asenapine — 5 or 10 mg BID
  Arms: Asenapine/Asenapine
Drug: Asenapine — 5 or 10 mg BID
  Arms: Placebo/Asenapine

SUMMARY:
Schizophrenia is a brain disease. The primary features of schizophrenia are characterized by Positive symptoms (symptoms that should not be there, inability to think clearly, to distinguish reality from fantasy i.e., hearing voices) and Negative symptoms (a reduction or absence of normal behaviors or emotions, i.e., unable to manage emotions, make decisions and relate to others). Other symptoms include reduced ability to recall and learn new information, difficulty with problem solving, or maintaining productive employment. The symptoms of schizophrenia may be due to an imbalance in chemicals in the brain, primarily dopamine and serotonin, which enables brain cells to communicate with each other.

The clinical development of asenapine, as described in the 2007 IDB appears to have antipsychotic activity with superior symptomatic control compared to placebo and an improved safety profile compared to currently available neuroleptics. Its fast dissolving formulation may further add to treatment compliance. While various titration schedules have been used in previous studies, dose increases at 5 mg BID (twice daily) up to 10 mg BID have been well tolerated. Therefore, further exploration in a larger group of subjects with acute exacerbation of schizophrenia using an asenapine flexible dosing design ( 5 or 10 mg BID) will mimic actual clinical practice in a long-term 52-week extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Completed the short-term 041023 trial (NCT00156104)
* Continued to meet all demographic and procedural inclusion criteria of the short-term trial upon entry into this long-term extension trial
* Sign a written informed consent for the 041513 trial.
* Demonstrated an acceptable degree of compliance with trial medication in the short-term trials in the opinion of the investigator

Exclusion Criteria:

* CGI-S (Clinical Global Impressions of Severity of Illness) score of greater than or equal to 6 (severely psychotic)
* Occurrence(s) of AEs (adverse events) or other clinically significant findings that would prohibit their continuation
* Met any of exclusion criteria regarding medical/psychiatric status listed in the 041023 short-term trial
* Met exclusion criteria for medication status in short-term trials except for antidepressants and mood stabilizers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Note that one participant in each of the Placebo/Asenapine and Asenapine/Asenapine groups was enrolled but did not receive treatment. Thus, the numbers who started the period will be greater than the numbers presented at baseline and for analysis.
Groups:
- Placebo/Asenapine: Placebo in Original Study (NCT00156104) and Asenapine 5 or 10 mg BID (twice daily) in Current Long-Term Extension
- Asenapine/Asenapine: Asenapine 5 or 10 mg BID in Original Study and in Current Long-Term Extension
- Haloperidol/Haloperidol: Haloperidol 2-8 mg BID in Original Study and in Current Long-Term Extension
Period: Overall Study
Arm/Group | Placebo/Asenapine | Asenapine/Asenapine | Haloperidol/Haloperidol
Started | 51 | 93 | 43
Completed | 20 | 30 | 16
Not Completed | 31 | 63 | 27
Not completed — Enrolled But Never Received Treatment | 1 | 1 | 0
Not completed — Adverse Event | 8 | 11 | 4
Not completed — Lack of Efficacy | 2 | 9 | 3
Not completed — Withdrawal by Subject | 13 | 26 | 16
Not completed — Lost to Follow-up | 5 | 7 | 1
Not completed — Other | 2 | 9 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Asenapine | Asenapine/Asenapine | Haloperidol/Haloperidol | Total
Number analyzed (Participants) | 50 | 92 | 43 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.6) | 35.3 (10.4) | 39.9 (11.6) | 38.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 37 | 25 | 84
  Male | 28 | 55 | 18 | 101

OUTCOME MEASURES:

1. Primary Outcome: Loss of Effect Over Time
Description: Loss of effect in subjects who had >=30% decrease from baseline in Positive and Negative Syndrome Scale (PANSS) score at the end of the original trial (NCT00156104) preceding the long-term extension.
  PANSS is a 30-item clinician-rated instrument for assessing symptoms of schizophrenia. Scores range from 30-210; higher scores indicate greater severity.
  Loss of effect = increase in total PANSS >=30% from start of current study; subjective worsening of schizophrenia/request for dose increase; Clinical Global Impressions of Severity of Illness score >=6; discontinuation for lack of efficacy.
Time Frame: Throughout the 52 weeks of the trial.
Population: These are participants who completed the original acute-phase trial (41023) with a decrease from baseline in Positive and Negative Syndrome Scale (PANSS) score >= 30%, received at least one dose in the current long-term extension, and had at least one post-baseline PANSS assessment during the extension.
Measure: Number; unit: Participants
Arm/Group | Placebo/Asenapine | Asenapine/Asenapine | Haloperidol/Haloperidol
Number analyzed (Participants) | 30 | 65 | 29
Participants
  <=Week 1 | 7 | 15 | 6
  >Week 1 to Week 2 | 3 | 4 | 4
  >Week 2 to Week 4 | 1 | 14 | 3
  >Week 4 to Week 8 | 3 | 3 | 1
  >Week 8 to Week 12 | 2 | 1 | 1
  >Week 12 to Week 16 | 3 | 1 | 4
  >Week 16 to Week 20 | 0 | 1 | 1
  >Week 20 to Week 24 | 0 | 3 | 0
  >Week 24 to Week 28 | 0 | 1 | 0
  >Week 28 to Week 32 | 1 | 3 | 1
  >Week 32 to Week 36 | 0 | 0 | 0
  >Week 36 to Week 40 | 0 | 0 | 1
  >Week 40 to Week 44 | 0 | 0 | 0
  >Week 44 to Week 48 | 0 | 0 | 0
  >Week 48 to Week 52 | 2 | 5 | 2
Statistical Analysis 1: Comparison: Placebo/Asenapine; Test type: Superiority or Other; Kaplan-Meier Estimate of Loss of Effect = 0.8619, 95% CI [0.6912 to 0.9644] — Loss of effect = increase in total PANSS >=30% from start of current study; subjective worsening of schizophrenia/request for dose increase; Clinical Global Impressions of Severity of Illness score >=6; discontinuation for lack of efficacy
Statistical Analysis 2: Comparison: Asenapine/Asenapine; Test type: Superiority or Other; Kaplan-Meier Estimate of Loss of Effect = 0.8834, 95% CI [0.7744 to 0.9550] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Haloperidol/Haloperidol; Test type: Superiority or Other; Kaplan-Meier Estimate of Loss of Effect = 0.9376, 95% CI [0.7631 to 0.9952] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Median Survival Time of Effect
Description: Kaplan-Meier estimate of median time to loss of effect in subjects who had >=30% decrease from baseline in PANSS score at the end of the original trial (NCT00156104) preceding the long-term extension.
  PANSS is a 30-item clinician-rated instrument for assessing symptoms of schizophrenia. Scores range from 30-210; higher scores indicate greater severity.
  Loss of effect = increase in total PANSS >=30% from start of current study; subjective worsening of schizophrenia/request for dose increase; Clinical Global Impressions of Severity of Illness score >=6; discontinuation for lack of efficacy.
Time Frame: 52 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo/Asenapine | Asenapine/Asenapine | Haloperidol/Haloperidol
Number analyzed (Participants) | 30 | 65 | 29
Days | 57 [15 to 111] | 31 [28 to 140] | 85 [15 to 118]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored continually through 52 weeks of treatment and 1 month of posttreatment follow-up.
Description: Information regarding AEs was obtained by questioning or examining the subject at each visit, and recording complaints and symptoms. Reports are for all serious AEs and treatment-emergent nonserious AEs.
Arm/Group | Placebo/Asenapine | Asenapine/Asenapine | Haloperidol/Haloperidol
Serious Adverse Events (participants affected / at risk) | 12/50 | 13/92 | 6/43
Other Adverse Events (participants affected / at risk) | 28/50 | 54/92 | 25/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Asenapine (N=50) | Asenapine/Asenapine (N=92) | Haloperidol/Haloperidol (N=43)
DRUG EXPOSURE DURING PREGNANCY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HYPONATREMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
SCHIZOPHRENIA (Psychiatric disorders) | 7 (8) | 8 (14) | 5 (6)
SCHIZOPHRENIA, PARANOID TYPE (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ABORTION INDUCED (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Asenapine (N=50) | Asenapine/Asenapine (N=92) | Haloperidol/Haloperidol (N=43)
CONSTIPATION (Gastrointestinal disorders) | 4 (5) | 4 (4) | 3 (3)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 3 (3) | 2 (2) | 6 (6)
VOMITING (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (4)
ASTHENIA (General disorders) | 5 (10) | 7 (8) | 6 (6)
INFLUENZA (Infections and infestations) | 3 (3) | 4 (4) | 3 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 6 (6) | 1 (1)
WEIGHT DECREASED (Investigations) | 2 (2) | 5 (6) | 0 (0)
WEIGHT INCREASED (Investigations) | 1 (1) | 3 (3) | 3 (3)
AKATHISIA (Nervous system disorders) | 4 (6) | 6 (7) | 3 (5)
DIZZINESS (Nervous system disorders) | 3 (3) | 2 (4) | 1 (1)
HEADACHE (Nervous system disorders) | 9 (17) | 10 (13) | 7 (8)
PARKINSONISM (Nervous system disorders) | 3 (3) | 10 (14) | 3 (7)
SOMNOLENCE (Nervous system disorders) | 5 (5) | 4 (6) | 1 (1)
TREMOR (Nervous system disorders) | 2 (3) | 3 (3) | 4 (6)
AGITATION (Psychiatric disorders) | 1 (2) | 7 (8) | 2 (3)
ANXIETY (Psychiatric disorders) | 3 (6) | 7 (12) | 2 (2)
DEPRESSION (Psychiatric disorders) | 1 (2) | 2 (2) | 3 (3)
INSOMNIA (Psychiatric disorders) | 12 (15) | 17 (34) | 4 (4)
SCHIZOPHRENIA (Psychiatric disorders) | 5 (5) | 9 (11) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Except for compelling legal reasons, neither the sponsor nor the investigator will communicate to third parties any result of the clinical trial before the CTR has been released by the sponsor.